CLINICAL TRIAL: NCT00578591
Title: CHIMERIC MONOCLONAL CD-20 ANTIBODY (RITUXIMAB) FOR STEROID REFRACTORY ACUTE GRAFT VERSUS HOST DISEASE (SR-AGVHD): A PILOT STUDY
Brief Title: Rituximab for GVHD
Acronym: Rituximab GVHD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No eligible patients were identified so the study was terminated.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rammurti Kamble, Principal Investigator, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19734; RITUXIMAB GVHD; NCT00624897 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Graft vs Host Disease; Alogenic Hematopoietic Transplant
Keywords: Graft Versus Host Disease; GVHD; allogeneic hematopoietic transplant; AHT; posttransplant; Rituximab
MeSH Terms: conditions — Graft vs Host Disease | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient (Experimental): Four Rituximab doses administered to patients who have developed SR-aGVHD following allogeneic hematopoietic transplant (AHT)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m^2 is given weekly X 4. For patients with a partial response, an additional 4 doses will be permitted as needed (after 4 weeks from the last dose).
  Diagnosis of grade II to IV aGVHD will be confirmed, whenever possible, by a biopsy taken from at least one of the following three sites: skin, gut, or liver.

SUMMARY:
This is a prospective, open-label pilot study in which 4 doses of Rituximab are administered to patients who have developed SR-aGVHD following allogeneic hematopoietic transplant (AHT). The study is designed to determine the overall survival at 180 days after treatment with rituximab, and evaluates the safety and clinical response to rituximab in this study population. Study entry: Patients must enter study on or before day +100 posttransplant.

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGVHD), one of the most important complications of allogeneic hematopoietic stem cell transplantation (HSCT) is associated with significant morbidity and mortality. Grades II to IV aGVHD occur in 30% to 50% of matched related donor recipients and 50% to 70% of unrelated donor recipients. Standard first-line treatment consists of methylprednisolone at a dose of 2 mg/kg/d or equivalent that produces response rates of 63% to 95% for grade II, 17% to 39% for grade III, and 0% to 6% for grade IV aGVHD. In aggregate, approximately 40% to 50% of patients with acute GVHD experience a complete or partial response with primary therapy, whereas 20% to 60% require salvage treatments. The 1994 consensus conference on acute GVHD grading reported 100-day survival rates of 78% to 90% with grade I, 66% to 92% with grade II, 29% to 62% for grade III, and 23% to 25% for grade IV. The higher mortality rates were directly attributable to acute GVHD or to the subsequent immunosuppression from high-dose corticosteroids and other medications required for treatment of GVHD.

Despite several studies seeking to improve first-line therapy for acute GVHD, standard care remains moderate-dose corticosteroids. Higher initial doses of corticosteroids, a more prolonged steroid tapering course, and addition of murine or equine anti-T-cell antibodies to standard GVHD therapy all failed to improve response rates. Acute GVHD therefore remains an unfavorable complication of transplantation that is difficult to manage. Various immunosuppressants including, Anti-thimocyte globulin (ATG), Denileukin Diftitox, Mycophenolate mofetil, Pentostatin, Infliximab, Rapamycin, Inolimomab and Daclizumab have been tried with variable success (table-1 in full protocol); there remains no consensus on the second-line treatment of aGVHD.

Acute graft-versus-host-disease (aGVHD) is mediated by donor T-cells. The preventative and therapeutic strategies described above have therefore focused on quantitative reduction in T cells or reduction of their function through immune-modulation. The role of B-lymphocytes in the pathogenesis of GHVD is unclear. Recent reports of successful use of rituximab in cGVHD support the hypothesis that a coordinated B and T cell response is instrumental in cGVHD. The significance of B-cells in pathogenesis of aGVHD is unknown.

Steroid Refractory Acute Graft-Versus-Host-Disease (SR-aGVHD) Initial treatment for aGVHD routinely consists of intensifying the dose of corticosteroids. This condition is called steroid-resistant (SR) aGVHD and requires secondary intervention.

Rituximab is a human/murine chimeric monoclonal anti CD-20 antibody that is extensively used in patients with B-cell non-Hodgkin's lymphoma, or with autoimmune disease. The incidental observation of improvement in aGVHD following rituximab infusion for transplant-associated thrombotic thrombocytopenic purpura (TA-TTP) and subsequent complete resolution of multi-agent refractory aGVHD in two patients forms the basis of this proposed pilot study. Table-2 (in full protocol) describes the patients and their responses to rituximab at our own institution.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute graft-versus-host disease (aGVHD)
2. Steroid-refractory aGVHD with any of the following: a) No change in the stage of skin aGVHD after 1 week of 2 mg/kg per day or more methylprednisolone. b) Progression of acute GVHD (ie, increase in disease stage by at least 1) of skin GVHD or lack of response of visceral (liver, GI) aGVHD despite treatment with 2 mg/kg per day or more methylprednisolone for at least 72 hours. c) Progression of visceral aGVHD despite treatment with 2 mg/kg per day or more methylprednisolone for at least 48 hours d) Visceral aGVHD progressing to stage 4 after 24 hours of 2 mg/kg per day or more methylprednisolone.
3. Grade II-IV aGVHD requiring systemic therapy within 24-48 hours of diagnosis. Biopsy confirmation of aGVHD is strongly recommended but not required; enrollment should not be delayed awaiting biopsy or pathology results.
4. Patients must have received corticosteroids at greater than or equal to 2 mg/kg/day for a minimum of 72 hours prior to study entry (first-line aGVHD treatment).
5. ANC greater than 500/uL x 3 days (must have evidence of engraftment).
6. Patient is <100 days posttransplant
7. Any age, sex, ethnicity.
8. Karnofsky score/Lansky score of greater than 20
9. Men and women of child-bearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) for the duration of the study and should continue such precautions for 6 months after receiving the study drug infusion.
10. Parent(s)/legal guardian must give informed consent.

Exclusion Criteria:

1. Chronic GVHD (defined as GVHD occurring beyond 100 days of the hematopoietic transplant).
2. Isolated upper gastrointestinal GVHD as sole manifestation of acute GVHD.
3. Isolated grade I or II skin GVHD as sole manifestation of aGVHD.
4. GVHD following donor lymphocyte infusion (DLI).
5. Other investigational agents for the treatment or prophylaxis of GVHD within the past 2 weeks. An investigational drug is defined as one that is being given on study, requiring informed consent.
6. Use of rituximab in the conditioning regimen for hematopoietic transplant.
7. Prophylactic immunosuppression tapered or stopped for treatment of leukemia relapse or minimal residual disease.
8. Patients with uncontrolled infection(s) i.e. documented bacterial, viral or fungal infection within 72 hours prior to study entry. Neither continuation of antibiotics for a controlled infection nor prophylactic/empiric antibiotics warrant exclusion. Patients with a C. difficile infection will not be excluded.
9. Patients with any one of the following opportunistic infections documented within 8 weeks prior to study entry are excluded: pneumocystis carinii, aspergillosis, histoplasmosis, atypical mycobacterium infection or other pathogenic molds/fungi.
10. Patients with hypotension believed to be secondary to sepsis syndrome or heart failure requiring > 1 inotropic agent, or dopamine >5mcg/kg/minute for blood pressure support.
11. Mechanical ventilatory support.
12. Relapsed, refractory, or second malignancies at the time of study entry.
13. Previous grade IV severe adverse reaction to rituximab.
14. Any allergy to murine products.
15. Documented HIV or HBV infection.
16. Patients with grade IV renal, hepatic, pulmonary, or neurologic toxicity by National Cancer Institute (NCI) Common Toxicity Criteria (CTC). 17. Patients with history of congestive heart failure, defined as cardiac dysfunction requiring inotropic support other than dopamine at <= 5mcg/kg/minute.

18. Autologous or syngeneic transplants.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Complete response rate at 4 and 8 weeks in patients with SR-GVHD treated with Rituximab. | 2 months

SECONDARY OUTCOMES:
Survival at day 180 after txt with rituximab. | 6 months
Partial response rates at 4 weeks and 8 weeks, mixed response rate, and disease progression in patients treated with these regimens. | 2 months
Treatment failure rate at 2 weeks (no response, progression, or mortality). | 2 weeks
Safety of rituximab in SR-GVHD | 2 years
Time to aGVHD improvement. | 2 years
Incidence of GVHD flares requiring further therapeutic intervention within 90 days of therapy. | 3 months
Incidence of discontinuation of immune suppression without flare by days 90, 180, and 270 post therapy. | 9 months
Incidence of chronic GVHD by 9 months (Day 270) | 9 months
Measurement of total dose of steroids. | 1 year
Overall survival at 6, 9 and 12-month post initiation of therapy. | 1 year
Incidence of systemic infections within 3 months of initiation of therapy. | 3 months
Relapse of primary disease. | 2 years
- Changes in the Karnofsky/Lansky performance status. - Incidence of Epstein-Barr virus-associated lymphoma - Recovery of T-and B-cells. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rammurti Kamble, MD, Principal Investigator — Baylor College of Medicine/TCH/Methodist
Locations (2):
- United States (2):
  - Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas